CLINICAL TRIAL: NCT02425345
Title: Women's Health Initiative Strong and Healthy Study
Acronym: WHISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of California, San Diego (Other); Stanford University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4R33HL151885-02 (NIH); 1U01HL122280-01A1 (NIH); 1U01HL122273-01A1 (NIH); RG1001184 (Other: Fred Hutchinson Cancer Center)
Record Dates: First submitted 2015-04-16; First posted 2015-04-24 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Infarction; Stroke; Cardiovascular Mortality; Hip Fractures; Falls; Mortality; Venous Thromboembolic Event; Peripheral Artery Disease; Physical Function; Coronary Revascularization; Mobility and Independence; Clinical (Non-hip) Fractures; Sleep; Depressive Symptoms
Keywords: Physical Activity; National Institute of Aging Go4Life; Postmenopausal Women; Balance; Strength; Exercise; Cardiovascular Disease; Stroke; Mortality; Myocardial Infarction; Falls; Venous Thromboembolic Event; Peripheral Artery Disease; Physical Function; Mobility and Independence; Coronary Artery Bypass Graft (CABG); Percutaneous Coronary Intervention (PCI); Hip Fractures; Cardiovascular Mortality; Clinical (non-hip) Fractures; Sleep; Depressive Symptoms
MeSH Terms: conditions — Myocardial Infarction; Stroke; Hip Fractures; Peripheral Arterial Disease; Fractures, Bone; Depression; Motor Activity; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Activity Intervention (Experimental): The Physical Activity Intervention Group will receive guidance on being physically active, including aerobics, flexibility, balance, strength, and decreased sedentary time. The primary resource is the National Institute of Aging Go4Life exercise and physical activity materials. The materials are based on the United States national guidelines for physical activity for older adults
  Interventions: Behavioral: Physical Activity
- Usual Activity Control (No Intervention): Usual activity

INTERVENTIONS:
Behavioral: Physical Activity — The PA intervention will consist of a multimodal activity program of aerobics, balance, strength, flexibility. The intervention will involve encouraging participants to increase all forms of PA throughout the day and to decrease sedentary time, such as sitting. This may include activities such as leisure sports, gardening, use of stairs instead of escalators, leisurely walks with friends, and less use of remote control devices.The intervention is conducted primarily by mail with website support and resources available.
  Arms: Physical Activity Intervention

SUMMARY:
The WHISH trial applies state-of-the science behavioral principles and currently available technologies to deliver a physical activity intervention without face-to-face contact to ~25,000 older U.S. women expected to consent. It includes the National Institute of Aging (NIA) Go4Life® Exercise & Physical Activity materials 3 and WHISH developed targeted materials based on Go4Life® to provide inspirational tips and recommendations about how to achieve nationally recommended levels of PA and overcome barriers to exercise, with a means for self-monitoring and setting personal goals. The intervention builds upon evidence-based behavioral science principles and intervention components that have proven to be effective in increasing PA in older women, with innovative adaptive approaches to tailoring the delivery to meet individual (personal) needs.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in the Women's Health Initiative (WHI) Extension Study
* Known to be alive
* Cardiovascular outcomes will be available (enrolled in the WHI Medical Records Cohort or linked to Medicare Data)

Exclusion Criteria:

* Inability to walk
* Dementia
* Residing in a nursing home

Ages: 66 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 49331 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Events (Composite Myocardial Infarction, Stroke, Cardiovascular Mortality | 9 years
  Adjudicated events
Physical Function (Physical Function Score from self-report, RAND-36) | 9 years
  Rand-36 Physical Function Scale. Score 0-100; a higher score indicates a more favorable health state in regards to physical functioning.
Non-Cardiovascular Disease Mortality | 9 years
  Safety; adjudicated event
Hip Fracture | 9 years
  Safety; adjudicated event
Clinical (non-hip) Fracture | 9 years
  Safety
Falls | 9 years
  Safety; self-report

SECONDARY OUTCOMES:
Venous Thromboembolic Event | 9 years
  Adjudicated event
Peripheral Artery Disease | 9 years
  Adjudicated event
Mobility and Independence (Physical Function Score from self-report) | 9 years
  Self-report of ability to climb one flight of stairs or ability to walk one block. Scored 1, 2 or 3 with 1=limited a lot, 2=limited a little, 3=not limited at all. Either stairs or walk with score of 2 or 3 is defined as being able to be mobile.
Coronary Revascularization (Coronary Artery Bypass Graft or Percutaneous Coronary Intervention) | 9 years
  Safety; adjudicated events
Short Physical Performance Battery (SPPB) | 4 years
  Short Performance Battery (SPPB). Scoring uses the Look AHEAD methods that were based on Health ABC (Simonsick EM, Newman AB, Nevitt MC, et al. Measuring higher level physical function in well-functioning older adults: expanding familiar approaches in the Health ABC Study. J Gerontol Med Sci. 2001;56A,M644-M649.) The SPPB score is sum of three ratios, the Standing Balance Ratio (SBRatio), the Chair Stand Ratio (CSRatio), and the Usual Walk Ratio (UWRatio). The results are in a continuous score ranging from 0 to 3. s (balance, gait speed, stair stand) are each scored 0 or 1 with the three scores summed for an SPPB score of 0 to 3 from lowest to highest physical function. Implemented in a subset.
Sleep Disturbance | 4 years
  Self-report of sleep patterns such as falling asleep, waking during the night, quality of night's sleep. Score scale: 0 - 20; a higher score indicates greater sleep disturbance. Levine DW, Kaplan RM, Kripke DF, Naughton MJ, Shumaker SA. Factor structure and measurement invariance of the Women's Health Initiative Insomnia Rating Scale. Psycho Assess. 2003 Jun; 15(2):123-36.
Depressive Symptoms | 4 years
  Shortened version of the Center for Epidemiological Studies Depression Scale (CES- D). Score (probability) for depression. Score scale: 0 - 1; a higher score indicates a greater likelihood of depression. Burman M, Wells K, Leake B, Landsverk J. Development of a brief screening instrument for detecting depressive disorders. Medical care 1988; 26: 8, 775-789.

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Kooperberg, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Andrea Z LaCroix, PhD, Principal Investigator — University of California, San Diego; Marcia L Stefanick, PhD, Principal Investigator — Stanford University

REFERENCES:
- [Background] Stefanick ML, King AC, Mackey S, Tinker LF, Hlatky MA, LaMonte MJ, Bellettiere J, Larson JC, Anderson G, Kooperberg CL, LaCroix AZ. Women's Health Initiative Strong and Healthy Pragmatic Physical Activity Intervention Trial for Cardiovascular Disease Prevention: Design and Baseline Characteristics. J Gerontol A Biol Sci Med Sci. 2021 Mar 31;76(4):725-734. doi: 10.1093/gerona/glaa325. PMID 33433559
- [Derived] Mendoza-Vasconez AS, King AC, Chandler G, Mackey S, Follis S, Stefanick ML. Engagement With Remote Delivery Channels in a Physical Activity Intervention for Senior Women in the US. Am J Health Promot. 2024 Jun;38(5):692-703. doi: 10.1177/08901171241229537. Epub 2024 Feb 12. PMID 38344760
- [Derived] Stefanick ML, Kooperberg C, LaCroix AZ. Women's Health Initiative Strong and Healthy (WHISH): A pragmatic physical activity intervention trial for cardiovascular disease prevention. Contemp Clin Trials. 2022 Aug;119:106815. doi: 10.1016/j.cct.2022.106815. Epub 2022 Jun 9. PMID 35691486
- See also: Women's Health Initiative Strong and Healthy Pragmatic Physical Activity Intervention Trial for Cardiovascular Disease Prevention: Design and Baseline Characteristics — https://pubmed.ncbi.nlm.nih.gov/33433559/